CLINICAL TRIAL: NCT06378814
Title: Randomized Clinical Trial of Treatment Outcomes of Selective Versus Nonselective Caries Removal in Deep Carious Lesions in Permanent Teeth.
Brief Title: Outcome of Selective & Nonselective Caries Removal in Permanent Teeth
Acronym: RCT-SNCR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS N335444
Record Dates: First submitted 2024-03-12; First posted 2024-04-23 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Deep Caries; Carious Exposure of Pulp

STUDY DESIGN:
Intervention Model Description: two arms parallel randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Caries Removal (Experimental): This process will be conducted under an operating microscope to ensure precise removal of carious dentin on cavity walls. Only disorganized carious dentin on the cavity floor will be removed using hand instruments in the control group which is SCR group
  Interventions: Procedure: Selective Caries Removal (No Pulp Exposure); Procedure: Partial Pulpotomy (Pulp Exposed)
- Non selective caries removal (Experimental): On the other hand, removal of carious dentin on cavity floor will be completely up to hard sound dentine in NSCR group.
  Interventions: Procedure: Non-Selective Caries Removal (No Pulp exposure); Procedure: Partial Pulpotomy (Pulp Exposed)

INTERVENTIONS:
Procedure: Selective Caries Removal (No Pulp Exposure) — Caries excavation technique where clinician leaves carious tissue so close to pulp
  Other Names: SCR
  Arms: Selective Caries Removal
Procedure: Non-Selective Caries Removal (No Pulp exposure) — Complete caries removal even in areas so close to pulp
  Other Names: NSCR
  Arms: Non selective caries removal
Procedure: Partial Pulpotomy (Pulp Exposed) — In caes of Pulp exposure Amputation of inflamed coronal pulp and capping of remaining vital tissue
  Other Names: Miniature Pulpotomy

SUMMARY:
Patients presenting with deep decay within permanent teeth presents a common clinical challenge to dentists. The aim of this trial is to compare the success rate of the non-selective caries removal (NSCR) and selective caries removal (SCR) in managing deep caries, as both methods are commonly used in clinical practice.

This study will be a randomized controlled trial, with participants divided into two groups: NSCR group and SCR group. Participants of deep caries lesions (reaching more than two-thirds of dentin on periapical radiographs) Both groups will undergo either NSCR or SCR, followed by Partial Pulpotomy (PP) in cases with pulp exposure. Success rates will be assessed at follow-up visits scheduled 1, 3, and 5 years radiographs will be used to assess for pulp health(vitality).

The success rate of the two categories will be assessed using a scale that includes factors such as tooth vitality, caries recurrence, and clinical signs of pulpitis. The scale will be applied at follow-up visits. The trial will be conducted in post-graduate dental clinics at Guy's hospital.

Deep caries in permanent teeth is a common clinical problem that can lead to pulp exposure and subsequent restorative challenges. The aim of this study is to provide evidence-based guidance for clinicians in managing deep caries lesions, as both NSCR and SCR are commonly used in clinical practice. The results of this study will help clinicians to make informed decisions when choosing the appropriate treatment approach for their patients.

In conclusion, this trial aims to compare the success rate of NSCR and SCR in managing deep caries lesions in permanent teeth, as both methods are commonly used in clinical practice. The results of this study will provide valuable insights into the effectiveness of these two treatment approaches and will help clinicians to make informed decisions when choosing the appropriate treatment approaches.

DETAILED DESCRIPTION:
The clinical trial aims to compare the outcomes of non-selective versus selective caries removal.

1. Recruiting patients This will involve symptomatic patients attending Guy's and St Thomas's NHS Foundation Trust (GSTT) dental clinics. To ensure voluntary participation, potential volunteers will be informed that they are free to decline without providing a reason, with written informed consent gained. The study will assess the success and survival rates of different caries excavation techniques in common clinical use currently.

   Both techniques are used routinely as a standard of care at GSTT. Patients will receive the same treatment as caries removal, but the difference will be in the technique that will be used and the decision of which will be used will be by the randomization. Patients will be randomized on the base of the tooth to one of the two caries removal techniques.

   Competent, adult patients meeting inclusion criteria will receive appropriate dental care as part of their routine clinical management, and any abnormal findings will be communicated to them. Participants will be informed about the exposure to radiation involved in the study protocol and will receive periapical and bitewing radiograph. Periapical and bitewing radiographs are x rays those used routinely at GSTT. Also they will be informed that In the unlikely event of treatment failure, patients will be offered root canal treatment to provide definite care. Patients will be randomized through an audited clinical trials tool.
2. Clinical examination and treatment Any abnormal clinical findings identified as a result of participation in this study will be communicated to the participants, and they will receive appropriate dental care as part of their routine clinical management. If required, patients may be referred to the appropriate clinical team or clinician for treatment as appropriate. This includes clinicians in the dental hospital and/or medical practitioners. Participants will be informed of this in the patient information sheet and provide their consent. In the unlikely event of treatment failure, patients will be offered root canal treatment to provide definite care.
3. Biological samples, including dentin, saliva, oral swabs, and blood, will be acquired during restorative procedures and stored at -80°C for optimal preservation. Proteomic analysis will be performed using high-resolution liquid chromatography-tandem mass spectrometry (LC-MS/MS) on dentin and saliva samples, while enzyme assays will quantify protease activities, particularly focusing on matrix metalloproteinases (MMPs). Bacterial enumeration will be conducted using qPCR (Quantitative Polymerase Chain Reaction) techniques, offering both specificity and sensitivity in microbial identification, correlated with the microbial community composition as determined by sequencing approaches. Biological specimen will be obtained by trained, competent dentally-trained operators (trained post-graduate students who are treating patients routinely at Guy's clinics as they are part of dental team). Biological specimen will be stored and managed within HTA (Human Tissue Authorization)-approved freezers on site.

   PhD(Doctor of Philosophy) student is the involved with the samples transfer and analysis where she is going to take training and certificates needed including HTA certificate.
4. Radiation exposure will be limited to radiographs necessary in routine care. No extra radiation will be given to patients as they are all routine of care radiographs at GSTT.
5. Confidentiality will be ensured by Pseudo-anonymization which will be performed by assigning a code to the patient's ID (Identification) number. All data and decoding will be kept separately on two different password-protected computers at each site. Access to the decoded data will be restricted to the chief investigator and academic supervisors until interim or final statistical analysis. All patients will be assured confidentiality, and no data submitted to statistical analysis will be traceable back to an individual patient.

The clinical trial will adhere to the principles of the Declaration of Helsinki. Patients may withdraw from the study at any time, and their clinical care will be unaffected.

ELIGIBILITY:
Inclusion Criteria:

1. Dental patients from routine dental care at ADC (Acute Dental Care) clinics, both undergraduate and postgraduate dental clinics in Guy's Hospital.
2. Both male and female individuals aged 18 years and older.
3. Capable of providing informed consent.
4. Generally, in good overall health from a medical standpoint.
5. Possess at least one molar or premolar tooth exhibiting a clinically significant deep carious lesion, with or without carious pulp exposure.
6. Displaying signs and symptoms indicative of a normal pulp or reversible pulpitis.
7. positive response to the cold test (refrigerated gas).
8. Absence of spontaneous pain.
9. Absence of periapical lesions, as determined by routine radiographic examination

Exclusion Criteria:

1. Presence of fistulas or swelling.
2. Involvement of anterior teeth.
3. Evidence of external or internal root resorption.
4. Multiple teeth with carious lesions within the same quadrant.
5. Pregnancy in women.
6. Patients under the age of 18.
7. Individuals unable to provide informed consent.
8. Patients who have received antibiotics in the preceding month.
9. Immunocompromised patients.
10. Teeth with tooth surface loss resulting from traumatic parafunctional habits or teeth displaying craze lines.
11. Caries located beneath the gingival margin .
12. Teeth affected by periodontal issues, characterized by bone loss or severe gingival recession.
13. Teeth with pulp exposure where operators cannot achieve hemostasis after applying a cotton pellet soaked with 2.5% sodium hypochlorite (NaOCl) for three cycles, with each cycle consisting of a 2-minute application of NaOCl.
14. People with difficulty to understand the clinical trial concept, procedure and details including language barrier.
15. participants who are involved in other research at the same period of our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
To compare the success rate of maintaining pulp vitality assessed by pulp sensibility test between Selective Caries Removal or Non- Selective Caries Removal techniques after one year of the intervention. | After One year
  This study aims to compare between reported success rate (maintained pulp vitality) in cases of deep caries lesion when treated by by Selective caries removal and non-selective caries removal.
  Pulp sensibility tests will be used to assess the response of the pulp to external stimuli (pulp vitality).
  The success rate will be calculated as the ratio of cases with maintained pulp vitality to the total treated cases in each group.

SECONDARY OUTCOMES:
Periapical Health Assessment Using Periapical Index Score in Deep Caries Lesion Treatment | At 1, 3 and 5 years after the intervention
  The study aims to evaluate periapical health in the treatment of deep caries lesions using selective caries removal and partial pulpotomy. The assessment will be done using the Periapical Index Score. The Periapical Index Score is a standardized scoring system based on radiographic findings, allowing for the identification of healing or failure outcomes. The Periapical Index (PAI) score is a radiographic scale used in endodontics to evaluate the severity of periapical lesions. The scale ranges from 1 to 5, with higher scores indicating more severe periapical pathology. A score of 1 represents no changes, while a score of 5 indicates extensive destruction of periapical tissues. In summary, higher PAI scores correspond to worse outcomes, indicating greater periapical pathology, while lower scores reflect healthier periapical regions.
Quality of Life Assessment ( Using OHIP-14 questionnaire) in Deep Caries Lesion Treatment: A Comparative Study of Selective Caries Removal and Partial Pulpotomy | after one year of the intervention.
  This study aims to assess the impact of selective caries removal and partial pulpotomy on the quality of life of participants with deep caries lesions. Quantitative assessment will be done using the Oral Health Impact Profile-14 (OHIP-14). The Oral Health Impact Profile-14 (OHIP-14) is a questionnaire used to measure how oral health affects a person's quality of life. It consists of 14 items and assesses various aspects of oral health-related impact, such as physical discomfort, functional limitations, psychological discomfort, and social disability. The scores on the OHIP-14 range from 0 to 56, with higher scores indicating a greater negative impact on quality of life. In summary, higher OHIP-14 scores signify a worse outcome, indicating a higher burden of oral health problems and a greater impact on daily life functioning. Lower scores indicate a better outcome, reflecting a lesser impact of oral health issues on overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mannoci, Professor, Principal Investigator — professor of endodontics